CLINICAL TRIAL: NCT00755209
Title: Tranexamic Acid for Preventing Progressive Intracranial Haemorrhage in Adults With Traumatic Brain Injury; a Randomised, Double-blinded, Placebo-controlled Trial
Brief Title: Tranexamic Acid for Preventing Progressive Intracranial Haemorrhage in Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Thailand Research Fund (Other); Khon Kaen Hospital (Other Government)
Responsible Party: Principal Investigator, Surakrant Yutthakasemsunt, Dr., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE 510606
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Brain Injuries
Keywords: Traumatic brain injury (TBI); Adults; Moderately severe TBI; Delayed traumatic intracranial haemorrhage; Expanding traumatic intracranial haemorrhage; Progressive intracranial haemorrhage (PIH); Antifibrinolytic agent; Tranexamic acid (TXA); Randomised, placebo-controlled trial; Human
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transamin (Placebo Comparator): Drug: tranexamic acid
  Loading 1 gram (~20 mg/kg) 100cc solution infuses in 30 minutes Maintenance 1 gram (~2.5 mg/kg/hr) 1000cc solution infuses in 8 hours
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — Loading 1 gram (~20 mg/kg) 100cc solution infuses in 30 minutes Maintenance 1 gram (~2.5 mg/kg/hr) 1000cc solution infuses in 8 hours
  Other Names: Transamin

SUMMARY:
The study's objective is to evaluate the effectiveness and safety of tranexamic acid for adult patients with moderate to severe TBI.With the research question as "Does TXA reduce the incidence of progressive intracranial haemorrhage by 50% compared to placebo in moderate to severe adult TBI patients at Khon Kaen Hospital?"

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a major public health problem with poor outcome especially with progressive intracranial haemorrhage (PIH) in severe patients. There are links between coagulopathic change after brain injury and delayed traumatic haemorrhage revealed by CT brain. Antifibrinolytic treatment can reduce blood loss after surgery and perhaps in moderate to severe TBI by similar haemostatic responses. It is justified to determine benefit for reversing hyperfibrinolysis after TBI. Tranexamic acid (TXA) has been shown to have significant clinical benefit in effectively reducing surgical bleeding in systematic reviews. It has been shown to have no effect on coagulation parameters and no demonstrated harmful effect in systematic reviews. This study is designed to determine the effectiveness of TXA in preventing PIH in patients with moderate to severe TBI. The treatment regimen if effective can be applied in general trauma practice worldwide.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe injuries(post-resuscitation scores GCS 4-12)
* age >= 16 year
* non-penetrating TBI in 8 hours onset
* first CT brain in 8 hours onset
* non neurosurgical OR in 8 hours onset

Exclusion Criteria:

* patients with coagulopathy
* serum creatinine over than 2 mg%
* with associated major organ injury requiring surgery within 8 hours of injury
* pregnancy
* receiving any medication which affects haemostasis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Progressive intracranial haemorrhage at 24 ± 8 hours confirmed by repeated CT Brain | 24 ± 8 hours

SECONDARY OUTCOMES:
Functional scale (GOS), mortality, operative treatment (later surgery for bleeding), adverse effect and transfusion need | at discharge period

CONTACTS AND LOCATIONS:
Overall Officials: Surakrant - Yutthakasemsunt, M.D., Study Chair — Faculty of Medicine; Khon Kaen University and Surgical unit; Khon Kaen Regional Hospital, Thailand; Warawut - Kittiwattanagul, M.D., Principal Investigator — Surgical Unit, Khon Kaen Regional Hospital, Thailand; Parnumas - Piyavechvirat, M.D., Principal Investigator — Surgical Unit, Khon Kaen Regional Hospital, Thailand; Professor Pisake - Lumbiganon, M.D.,M.S., Principal Investigator — Faculty of Medicine; Khon Kaen University, Thailand; Asso. Professor Bandit - Thinkhamrop, M.P.H., Ph.D, Principal Investigator — Faculty of Public Health; Khon Kaen University, Thailand; Professor Nakornchai - Phuenpathom, B.Sc., M.D., Principal Investigator — Faculty of Medicine, Prince of Songkla University, Thailand
Locations (1):
- Khon Kaen Regional hospital, Muang District, Changwat Khon Kaen, Thailand